CLINICAL TRIAL: NCT00487253
Title: Randomized Clinical Trial of the Efficacy and Tolerability of Oral Miltefosine Versus Parenteral Antimony for the Treatment of Pediatric Cutaneous Leishmaniasis in Colombia
Brief Title: Oral Miltefosine for the Treatment of Pediatric Cutaneous Leishmaniasis in Colombia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centro Internacional de Entrenamiento e Investigaciones Médicas (Other)
Collaborators: Instituto Colombiano para el Desarrollo de la Ciencia y la Tecnología (COLCIENCIAS) (Other Government); INS (Unknown); Instituto Nacional de Dermatología Centro dermatológico Federico Lleras Acosta (Unknown)
Responsible Party: Santiago Nicholls, Instituto Nacional de Salud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50100119
Record Dates: First submitted 2007-06-14; First posted 2007-06-18 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Cutaneous Leishmaniasis; Leishmania Viannia; Pediatric; Miltefosine; Randomized; Colombia
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — miltefosine; Meglumine Antimoniate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Oral administration of Miltefosine, doses: 1,5mg to 2,5mg/kg/day, during 28 days.
  presentation: capsulas 10mg and 50mg Miltefosine (Impavido®)
  Interventions: Drug: Miltefosine
- Group 2 (Active Comparator): Administration of Parenteral meglumine antimoniate, Glucantime® Amp 5ml (83mg/ml). Dosage:20mg/kg/day, during 20 days.
  Interventions: Drug: Meglumine antimoniate

INTERVENTIONS:
Drug: Miltefosine — Oral Miltefosine, dosage 1,5mg -2,5mg/kg/day, during 28 days.
  Other Names: Miltefosine cap 10mg and 50mg, Impavido® (Zentaris)
  Arms: Group 1
Drug: Meglumine antimoniate — Parenteral meglumine antimoniate Amp of 5ml (83mg/ml). Dosage: 20mg/kg/day one doses IM, during 20 days.
  Other Names: Glucantime® of Aventis: Amp of 5ml (83mg/ml).
  Arms: Group 2

SUMMARY:
The purpose of this randomized, open label clinical trial is to determine if oral miltefosine is a safe and effective alternative, compared with parenteral meglumine antimoniate for the treatment of pediatric Cutaneous caused by L. Viannia species in Colombia.

ELIGIBILITY:
Inclusion Criteria:

* 2 to 12 years of age (inclusive)
* Parasitologically confirmed CL
* Availability to receive supervised treatment for 28 days (i.e., directly observed therapy, to ensure the therapy is appropriately administered and received - e.g., the miltefosine is "swallowed")
* Availability to return for follow-up visits for at least 6 months after treatment is initiated

Exclusion Criteria:

* Weight under 10kg
* Previous use of SbV, miltefosine or other antileishmanial therapy
* Simultaneous mucosal lesions suggestive of or proven to be mucosal leishmaniasis
* If a girl, ability to reproduce (history of menarche)
* Relative or absolute contraindications for the use of SbV drugs or miltefosine, including history of cardiac, renal or hepatic disease
* Patients with pretreatment haemoglobin <10g/dl or blood urea nitrogen (BUN), serum creatinine, ALT, AST or amylase values that exceed the upper limit of normal
* If living in Malaria endemic areas (eg. Tumaco) only: A positive malaria thick smear

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2007-07; Primary Completion 2010-02 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be the proportion of "Therapeutic Failures" diagnosed during the final (week 26) visit or before, according to defined clinical criteria. | 26 weeks (6 months)
Evidence of clinical or laboratory toxicity during the treatment period. | During the treatment period (20 or 28 days)

SECONDARY OUTCOMES:
Proportion of patients with "parasitologic" response 26 weeks after the initiation of treatment. | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Luisa Consuelo Rubiano, MD, MSc, Principal Investigator — Centro Internacional de Entrenamiento e Investigaciones Médicas

REFERENCES:
- [Derived] Castro MDM, Cossio A, Velasco C, Osorio L. Risk factors for therapeutic failure to meglumine antimoniate and miltefosine in adults and children with cutaneous leishmaniasis in Colombia: A cohort study. PLoS Negl Trop Dis. 2017 Apr 5;11(4):e0005515. doi: 10.1371/journal.pntd.0005515. eCollection 2017 Apr. PMID 28379954
- [Derived] Rubiano LC, Miranda MC, Muvdi Arenas S, Montero LM, Rodriguez-Barraquer I, Garcerant D, Prager M, Osorio L, Rojas MX, Perez M, Nicholls RS, Gore Saravia N. Noninferiority of miltefosine versus meglumine antimoniate for cutaneous leishmaniasis in children. J Infect Dis. 2012 Feb 15;205(4):684-92. doi: 10.1093/infdis/jir816. Epub 2012 Jan 11. PMID 22238470